CLINICAL TRIAL: NCT02212145
Title: Long-term Follow-up of an Individual and Population-based Program Aimed at Preventing Cardiovascular Disease in Sollentuna Municipality
Brief Title: Follow-up of Sollentuna Prevention Program
Acronym: SoPP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Heart Lung Foundation (Other)
Responsible Party: Principal Investigator, Mai-Lis Hellénius, Professor, Professor, Karolinska Institutet
Other Study IDs: 20100473; 2012/1172-31/1 (Other: Regional Ethical Review Board, Stockholm)
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Cardiovascular Diseases
Keywords: prevention; cardiovascular disease; risk factors
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Screened group: Screened group is defined as those individuals who were willing to participate in the cardiovascular prevention program and all the individuals who lived in Sollentuna during the intervention.
- Relatives to the screened group: Relatives to individuals included in the screened group, who lived in Stockholm County at least during one year at the time of the intervention.
- Control group: Matched "controls" is going to be selected randomly from the population of Stockholm County minus Sollentuna Municipality with relevant background factors. The whole population will be used as a comparison group when evaluating the result from all the municipality of Sollentuna during 1988-1993.

SUMMARY:
To evaluate long-term effects of one individual- and population-oriented cardiovascular prevention programs in primary care.

DETAILED DESCRIPTION:
In Sweden there are unique opportunities to create a relevant comparison group for this study, which is of great importance to the value of this cohort study.

Of the three study populations two (2-3)will be created by using national registries.

1. The screened group consists of the individuals (n = 5938) who had direct contact with the prevention program, ie undergone a voluntary opportunistic cardiovascular screening (questionnaire, physical examination and testing in connection with visits to health centers) and the rest of all individuals who lived in Sollentuna Municipality between 1988-1993.
2. Relatives of individuals included in the screened group who lived in Stockholm county at the time of the intervention will be identified by the use of the Medical Birth Register and the Multi-Generation Register. Family members are defined as parents, siblings and children and husband / wife to those in thescreened group and will be analyzed in the same way as those who participated in the intervention for risk of developing cardiovascular disease and cancer.
3. The comparison group consists of the entire population of Stockholm County minus Sollentuna 1988-93, taking into account population changes (migration, birth, death) during the period.

This three populations will be followed-up in national registries and databases

All subjects will be monitored for example disease history, socio-economics and biochemical risk factors presented below national registries and research databases. When all the matches of national registers and a local register (AMORIS)have been done the database will de-identified and anonymized data to be available for statistical processing.

ELIGIBILITY:
Inclusion Criteria in the risk intervention group:

* Individuals 15 years of age or more who visited three (four) health care centres in Sollentuna 1988-1993 were offered to participate in the prevention program

Exclusion Criteria in the screened intervention group:

* Age < 15 years

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. The screened group who participated in the cardiovascular prevention program:
     (n=5938) and the rest of the population in Sollentuna Municipality.
  2. To the screened group matched "controls" will be selected randomly from the population of Stockholm County minus Sollentuna. The population in Sollentuna will compared to the population of Stockholm County minus Sollentuna Municipality.
  3. Relatives of individuals included in the intervention group and who lived in Stockholm County at the time of the intervention will be identified by use of national registers.
Sampling Method: Non-Probability Sample
Enrollment: 1600000 (Estimated)
Dates: Start 1988-06; Primary Completion 2015-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and mortality in acute myocardial infarction, stroke, cardiovascular disease, and overall mortality, a twenty year follow-up of a prevention program. | 24 years
  Long term follow-up of a cardiovascular prevention program by using Swedish national patient registries

SECONDARY OUTCOMES:
A follow-up of drug treatment of diabetes, dyslipidemia and hypertension | 24 years
  By using the drug register in Sweden do a follow-up of drug treatment in the cohort

OTHER OUTCOMES:
Incidence and mortality in cancer | 24 years
  Incidence and mortality in cancer - a twenty year follow-up by using the swedish cancer register
Consumption of medical care overall and for different diagnostic groups | 24 years
  To study medical care consumption overall for different diagnostic groups by using different registers in Sweden
Health economic aspects | 24 years
  Health economic aspects such as
  1. health care consumption in total and for different diagnostic groups
  2. care costs
  3. impact on indirect costs (lost working years and sick leave)
  4. intervention cost will be studied
Time trends of morbidity and mortality in acute myocardial infarction, stroke, cardiovascular disease and total mortality | 24 years
  To study time trends of morbidity and mortality in acute myocardial infarction, stroke, cardiovascular disease and total mortality by use of National Swedish registries.

CONTACTS AND LOCATIONS:
Overall Officials: Gunilla Journath, PhD, Principal Investigator — Karolinska Institutet

REFERENCES:
- [Derived] Journath G, Hammar N, Elofsson S, Linnersjo A, Vikstrom M, Walldius G, Krakau I, Lindgren P, de Faire U, Hellenius ML. Time Trends in Incidence and Mortality of Acute Myocardial Infarction, and All-Cause Mortality following a Cardiovascular Prevention Program in Sweden. PLoS One. 2015 Nov 18;10(11):e0140201. doi: 10.1371/journal.pone.0140201. eCollection 2015. PMID 26580968